CLINICAL TRIAL: NCT04004767
Title: Trial Ready Cohort for the Prevention of Alzheimer's Dementia (TRC-PAD)
Brief Title: TRC-PAD Program: In-Clinic Trial-Ready Cohort
Acronym: TRC-PAD
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other); Alzheimer's Clinical Trials Consortium (Other); Brigham and Women's Hospital (Other); Cleveland Clinic Lou Ruvo Center for Brain Health (Unknown)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Other Study IDs: ATRI-004; R01AG053798 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Preclinical Alzheimer's Disease; Prodromal Alzheimer's Disease; Alzheimer Disease; Dementia
Keywords: Alzheimer's; Prevention; Observational; Trial-Ready Cohort
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TRC-PAD Cohort: Individuals identified as being at an increased risk for memory loss caused by Alzheimer's disease dementia. Determination of risk based on a number of factors including family history, performance on memory tests, genetic tests and biomarker tests.

SUMMARY:
The purpose of the TRC-PAD study is to develop a large, well-characterized, biomarker-confirmed, trial-ready cohort to facilitate rapid enrollment into AD prevention trials utilizing the APT Webstudy and subsequent referral to in-clinic evaluation and biomarker confirmation. Participants with known biomarker status may have direct referral to the Trial-Ready Cohort.

If you are interested in being selected for the TRC-PAD study, you should first enroll in the APT Webstudy (https://www.aptwebstudy.org/welcome).

DETAILED DESCRIPTION:
TRC-PAD study is short for the "Trial-Ready Cohort for the Prevention of Alzheimer's Dementia". The purpose of the TRC-PAD study is to find many people (also called a "cohort") who are interested in participating in clinical trials aimed at discovering treatments that will reduce the risk of developing Alzheimer's dementia. TRC-PAD will help researchers enroll participants into these trials quickly to allow new treatments to be discovered as soon as possible.

The TRC-PAD study is for individuals, age 50 and older, who may be at increased risk for memory loss caused by Alzheimer's disease. To join the TRC-PAD study, you first need to be invited to complete an in-person TRC-PAD visit.

How can I be invited to an in-person visit for TRC-PAD? Members of the Alzheimer Prevention Trials (APT) Webstudy complete online questionnaires and memory tests. The results of these tests will identify individuals as being eligible for an in-person TRC-PAD visit. If you are not enrolled in the APT Webstudy, you may be invited to an in-person visit for TRC-PAD because other tests or procedures you have had suggest you might be eligible to participate.

How might the TRC-PAD Study help researchers learn more about Alzheimer's disease dementia? Alzheimer's disease remains one of the most important medical conditions for which there is no treatment. Among the top ten causes of death, Alzheimer's disease is the only one that cannot be prevented, cured, or even slowed. To change this, researchers are conducting clinical trials to find new treatments. These trials need to study large numbers of individuals and follow participants over long periods of time. The goal of TRC-PAD is to identify individuals for these trials. TRC-PAD will find a group of people who may be "at-risk" for developing Alzheimer's dementia in the future and are appropriate for prevention trials.

How does TRC-PAD decide that I may have an increased risk for developing Alzheimer's dementia? A person's risk for developing Alzheimer's dementia is determined by a number of factors including family history, performance on memory tests, and biological tests called biomarkers. Biomarkers are measurements in parts of the body - like blood tests or brain scans - to help assess the presence of, or potential to develop, a disease.

If I decide to join TRC-PAD, what happens? Individuals in the TRC-PAD study will complete several assessments to see if they qualify to join the cohort. This will include biomarker testing (via Positron Emission Tomography (PET) brain scan or spinal fluid collection), tests of memory and thinking, questionnaires about daily functioning, mood and behavior, genetic testing and routine blood and urine tests. Individuals who are determined to eligible to enroll in TRC will come back to the clinic every 6 months for brief longitudinal follow-up visits with questionnaires and testing until that individual qualifies for a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated availability and willingness to comply with all study procedures until referred to a clinical trial
3. Age 50-85 (inclusive)
4. Global Clinical Dementia Rating (CDR) score of 0 or 0.5 and no diagnosis of dementia
5. Has a study partner that is willing to participate as a source of information and has at least weekly contact with the participant (contact can be in-person, via telephone or electronic communication). The study partner must have sufficient contact such that the investigator feels the study partner can provide meaningful information about the participant's daily function.
6. In good general health as evidenced by medical history
7. Adequate visual and auditory acuity to allow neuropsychological testing
8. Fluent in English or Spanish
9. For females who are not surgically sterile or post-menopausal by two years, receiving a Positron Emission Tomography (PET) scan for amyloid biomarker confirmation: negative pregnancy test prior to amyloid PET scan
10. Completed six grades of education or has a good work history
11. Evidence of elevated or intermediate (subthreshold) levels brain amyloid as assessed by central review of amyloid PET or cerebrospinal fluid (CSF) data. Prior amyloid testing results may be used with approval from the Coordinating Center.

Exclusion Criteria:

1. Treatment with an another anti-amyloid investigational anti-amyloid drug or other experimental intervention within 12 months. Use of aducanumab or other approved anti-amyloid treatments allowed if stable for at least 3 months.
2. Enrolled in another interventional clinical trial within the last 12 weeks
3. Any significant neurologic disease such as Alzheimer's disease dementia, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
4. Major depression, bipolar disorder as described in DSM-V within the past 1 year or psychotic features, agitation or behavioral problems within 3 months, which could lead to difficulty complying with the protocol
5. History of schizophrenia (DSM V criteria)
6. History of alcohol or substance abuse or dependence within the past 2 years (DSM V criteria)
7. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results, or the participant's ability to participate in the study.
8. History within the last 3 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment
9. Clinically significant abnormalities in B12 or thyroid function tests (TFTs) that might interfere with the study. A low B12 is exclusionary, unless follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant.
10. Clinically significant abnormalities in screening laboratories or ECG.
11. For participants undergoing CSF collection: a current blood clotting or bleeding disorder, or significantly abnormal PT or PTT at screening or if on anti-coagulation (e.g. warfarin)
12. Participants whom the Site PI deems to be otherwise ineligible.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AD biomarker confirmed individuals who may be at an increased risk for memory loss caused by Alzheimer's disease dementia. Individuals at highest risk within the APT Webstudy will be referred for an in-person TRC-PAD visit. Individuals with known biomarker status may qualify for a direct referral to the trial-ready cohort.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Enrollment into preclinical and prodromal AD clinical trials | 5 years

SECONDARY OUTCOMES:
Optimization of adaptive risk algorithm to predict risk of amyloid positivity | 5 years
  The TRC-PAD program aims to optimize an innovative, adaptive risk algorithm to efficiently identify the most appropriate trial participants. Once optimized, this algorithm will be able to select amyloid positive individuals (and eventually tau and other neurodegenerative biomarkers) with >75% accuracy, greatly reducing future costly biomarker screen fails.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aisen, MD, Principal Investigator — USC Alzheimer's Therapeutic Research Institute (ATRI); Reisa Sperling, MD, Principal Investigator — Brigham and Women's Hospital; Jeffrey Cummings, MD, Principal Investigator — Cleveland Clinic Lou Ruvo Center for Brain Health
Locations (45):
- United States (45):
  - University of Alabama, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Gonzalez MD & Aswad MD Health Services, Miami, Florida
  - Wien Center for Alzheimer's Disease, Miami Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research Orlando, Orlando, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Synexus Clinical Research, The Villages, The Villages, Florida
  - Charter Research, LLC, Winter Park, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Headlands Eastern MA LLC, Plymouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Roper St. Francis Hospital, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of North Texas Health Sciences Center, Fort Worth, Texas
  - National Clinical Research, Inc., Richmond, Virginia
  - University of Washington / Seattle Institute for Biomedical and Clinical Research, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Background] Amariglio RE, Donohue MC, Marshall GA, Rentz DM, Salmon DP, Ferris SH, Karantzoulis S, Aisen PS, Sperling RA; Alzheimer's Disease Cooperative Study. Tracking early decline in cognitive function in older individuals at risk for Alzheimer disease dementia: the Alzheimer's Disease Cooperative Study Cognitive Function Instrument. JAMA Neurol. 2015 Apr;72(4):446-54. doi: 10.1001/jamaneurol.2014.3375. PMID 25706191
- [Background] Mormino EC, Papp KV, Rentz DM, Donohue MC, Amariglio R, Quiroz YT, Chhatwal J, Marshall GA, Donovan N, Jackson J, Gatchel JR, Hanseeuw BJ, Schultz AP, Aisen PS, Johnson KA, Sperling RA. Early and late change on the preclinical Alzheimer's cognitive composite in clinically normal older individuals with elevated amyloid beta. Alzheimers Dement. 2017 Sep;13(9):1004-1012. doi: 10.1016/j.jalz.2017.01.018. Epub 2017 Feb 28. PMID 28253478
- See also: APT Webstudy — https://www.aptwebstudy.org/welcome
- See also: ATRI Studies — https://keck.usc.edu/atri/research/studies/
- See also: Alzheimer's Clinical Trials Consortium — https://www.actcinfo.org/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT04004767/Prot_SAP_000.pdf